CLINICAL TRIAL: NCT04131777
Title: Post-Market Optimization Study of the EMPOWER® RF Catheter to Ablate Soft Tissue Lesions in the Lung
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Broncus Medical Inc (Industry)
Collaborators: Uptake Medical Technology, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Protocol 46
Record Dates: First submitted 2019-10-09; First posted 2019-10-18 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Lung Diseases
MeSH Terms: conditions — Lung Diseases | interventions — Catheters

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fixed lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Roll-in: Initial patients enrolled until optimal RF algorithm is determined
  Interventions: Device: Radiofrequency (RF) catheter
- Optimized: Patients treated using optimal RF algorithm
  Interventions: Device: Radiofrequency (RF) catheter

INTERVENTIONS:
Device: Radiofrequency (RF) catheter — A catheter introduced into the lung lesion via a bronchoscope, used to deliver radiofrequency (RF) energy for the purpose of ablation
  Other Names: EMPOWER® RF Catheter

SUMMARY:
A post-market study to assess the performance and safety of a RF ablation catheter to bronchoscopically ablate lung lesions will be evaluated in patients with confirmed diagnosis of non-small cell lung cancer or metastatic lung lesions who are scheduled for surgical resection.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, multi-center, post-market study of bronchoscopic radio frequency (RF) ablation treatment malignant lung lesions prior to surgical resection. Up to 15 patients will be treated at the participating sites.

Patients identified for the study will have been scheduled for surgical resection as part of their treatment for lung lesions. The RF ablation procedure will be performed during a standard-of-care bronchoscopic procedure at minimum of 24 hours prior to resection. The patients exits the study following surgical resection. The resected tissue will undergo pathological evaluation for tissue viability.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at screening
2. Proven NSCLC or pulmonary metastases from extra-thoracic primary tumor
3. Eligible for standard of practice lung resection (pneumonectomy, lobectomy)
4. Tumor/lesion > 2cm along the major diameter with no visible necrosis
5. Signed informed consent form

Exclusion Criteria:

1. An implantable pacemaker, defibrillator, or other active implants
2. Any other severe or life-threatening comorbidity that could increase the risk associated with bronchoscopic RF ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with non-small cell lung cancer (NSCLC) and/or pulmonary metastases that are recommended for curative lung resection (pneumonectomy, lobectomy). Enrolled patients will have a microscopically confirmed malignancy, ensuring patients are surgical candidates.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Performance - maximum diameter of zone of thermal necrosis surrounding treated lesion | The interval between ablation and tissue resection for pathological analysis is a minimum of 24 hours, but the exact interval depends on the investigator's standard of care
  Maximum diameter (in mm) of ablation zone (thermal necrosis) surrounding treated lesion as measured in resected tissue by quantitative histopathological and gross pathological analysis
Performance - ability of the user and device to deliver ablative treatment in accordance with the catheter's Instructions for Use | Assessed at the time of the RF ablation procedure
  The ability of the ablation treatment to be delivered as per the Instructions for Use will be assessed using a binary categorical scale (yes/no)
Safety - Adverse events (AEs) and serious adverse events (SAEs) | AEs and SAEs related to the RF procedure/device will be reported for the interval beginning with the RF ablation procedure and ending with the surgical resection of the ablated lung tissueion
  The incidence of reported adverse events and serious adverse events related to the RF ablation procedure/device

CONTACTS AND LOCATIONS:
Overall Officials: Felix J Herth, MD, PhD, Principal Investigator — Heidelberg University
Locations (1):
- Thoraxklinik Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: No